CLINICAL TRIAL: NCT01353885
Title: Outcomes Following Anterior Approach to Total Hip Arthroplasty: A Multi-Centre Observational Cohort Study
Brief Title: Outcomes Following Anterior Approach to Total Hip Arthroplasty
Acronym: AAP
Status: Terminated | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: Depuy-05072
Record Dates: First submitted 2011-05-11; First posted 2011-05-16 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Osteoarthritis, Hip
Keywords: Primary Osteoarthritis, Hip; Total Hip Arthroplasty; Anterior Approach; Posterior Approach; Anterolateral Approach; Cohort Study; Outcomes, Complication Rate; Outcomes, Quality of Life
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Anterior Approach THA: 500 Patients will be included who have received a total hip arthroplasty using the Anterior Approach. The anterior approach to total hip arthroplasty refers to an internervous approach to the hip, where the incision is made from the middle of the iliac crest, then curved distally and laterally to the anterior superior iliac spine (Kelmanovich et al., 2003). To optimize feasibility and applicability of our results, we will not standardize the use of cemented components, the implant manufacturer, or the femoral head size. Surgeons will use the manufacturer specific guides for insertion of the total hip arthroplasty.
- Posterior Approach THA: 100 patients will be enrolled who have received a total hip arthroplasty using the posterior approach. The posterior approach is performed by making a curved incision posteriorly on the greater trochanter (Jolles & Bogoch, 2004). The fascia lata is then incised and the fibers of the gluteus maximus split using dissection (Jolles & Bogoch, 2004). To ensure the feasibility and applicability of our findings, we will not standardize the use of cemented components, the implant manufacturer, or the femoral head size used in the posterior approach.
- Anterolateral Approach THA: 100 patients will be enrolled who have had a total hip arthroplasty using the anterolateral approach. An anterolateral approach to THA utilizes an intermuscular approach by incising the patient posteriorly and distally to the anterior superior iliac spine, extending distally to the greater trochanter along the shaft of the femur (Kelmanovich et al., 2003). To optimize the feasibility and applicability of our results, the implant manufacturer, femoral head size or the use of cemented components will not be standardized in this study.

SUMMARY:
Osteoarthritis disables approximately 10% of people who are 60 years or older and compromises the quality of life of more than 20 million Americans every year. Osteoarthritis is caused by the breakdown of cartilage that lines the bones at your joints from daily wear and tear and results in pain and restricted function. Total hip arthroplasty (THA) or total hip replacement, is currently one of the most successful and cost-effective treatments used to eliminate pain and restore function in those suffering from osteoarthritis. There are multiple ways to perform a THA. The main difference between each type is the point of incision in relation to a muscle on the outer surface of your hip bone: gluteus medius. The incision performed can be anterior (in front of the muscle), anterolateral (in front and to the side of the muscle), or posterior (from the back). Each of these approaches has its own advantages and disadvantages, but there is no evidence available that makes one better than the other. The purpose of this study is to determine which of the three approaches to THA is the most effective. The main outcome that will determine the most effective approach is the functional ability of the patients included in this study at 52 weeks. The investigators will also compare whether the patient's: length of hospital stay, use of assistive devices, need for revision surgery, ability to return to work, ability to relieve pain, complication rate, and quality of life. The investigators hypothesize that the anterior approach will be the most effective approach in reducing the rate of post-operative complications after THA.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women who are 18 years of age or older.
2. Primary diagnosis of hip arthritis (radiographically and clinically).
3. Patients undergoing an unilateral THA.
4. Provision of informed consent by patient.

Exclusion Criteria:

1. Patients being managed with alternative approaches (other than anterior, anterolateral or posterior THA) will be excluded.
2. Patients undergoing a revision THA.
3. Patients undergoing a bilateral THA.
4. Patients with infection around the hip (soft tissue or bone).
5. Patients who have had previous major hip surgery (hip arthroscopy is permitted) or hardware implanted in their hip.
6. Patients who are currently enrolled in another surgical intervention trial.
7. Patient has cognitive or language barriers that would limit completion of quality of life, pain, and function questionnaires in English.
8. Anticipated problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women who are 18 years of age or older with a primary diagnosis of hip arthritis (radiographically and clinically). Patients must be undergoing an unilateral THA and have had no previous major hip surgery (hip arthroscopy is permitted) or hardware implanted in their hip.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Patient Functional Ability | 52 Weeks
  Measured by the Hip Disability and Osteoarthritis Outcome Score (HOOS) questionnaire.

SECONDARY OUTCOMES:
Technical Parameters | 1 day - measured during and post-operatively
  Length of Incision (cm), Blood Loss (mL), Fluoroscopy Time (s), Operative Time (Min)
Length of Hospital Stay | 4 weeks
  Duration of time patient is in hospital post-operatively.
Use of Assistive Device | 52 weeks
  Presence of an assistive device(s) provided to patients at discharge and the length of time it takes the patient to discard the assistive device(s).
Revision Surgery | 52 weeks
  Occurrence and type of revision surgery required (if any)
Ability to participate in sports activities | 52 weeks
  Subjectively reported.
Return to Work | 52 Weeks
  Measured by the Work Limitations Questionnaire (WLQ)- short form format
Complication Rate | 52 Weeks
  We will define complications in patients as a constellation of clinical symptoms and laboratory examinations. These will include (but are not limited to) both intraoperative and postoperative complications; More specifically, musculoskeletal, cardiovascular, psychological, neurological, genitourinary, and wound-related complications.
Pain | 52 Weeks
  Measured by the EuroQol-5d (EQ-5D) and Hip Disability and Osteoarthritis Outcome Score (HOOS) questionnaires.
Quality of Life | 52 Weeks
  Measured by the EuroQol-5d (EQ-5D) and Hip Disability and Osteoarthritis Outcome Score (HOOS) questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, PhD, FRCSC, Principal Investigator — McMaster University; Joel Matta, MD, Principal Investigator — St. Joseph's Health Centre Toronto
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Jolles BM, Bogoch ER. Surgical approach for total hip arthroplasty: direct lateral or posterior? J Rheumatol. 2004 Sep;31(9):1790-6. PMID 15338502
- [Background] Kelmanovich D, Parks ML, Sinha R, Macaulay W. Surgical approaches to total hip arthroplasty. J South Orthop Assoc. 2003 Summer;12(2):90-4. PMID 12882247